CLINICAL TRIAL: NCT02539212
Title: A Randomized Controlled Trial of Microwave and Radiofrequency Ablation in the Treatment of Early-stage Hepatocellular Carcinoma Meeting Milan Criteria
Brief Title: Comparison of Microwave and Radiofrequency Ablation for Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chair, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 939530
Record Dates: First submitted 2015-08-12; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: microwave; radiofrequency; ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microwave ablation (Active Comparator): microwave ablation
  Interventions: Device: microwave ablation
- radiofrequency ablation (Active Comparator): radiofrequency ablation
  Interventions: Device: radiofrequency ablation

INTERVENTIONS:
Device: microwave ablation — ultrasound-guided microwave ablation is performed to treat hepatocellular carcinoma patients
  Arms: microwave ablation
Device: radiofrequency ablation — ultrasound-guided radiofrequency ablation is performed to treat hepatocellular carcinoma patients
  Arms: radiofrequency ablation

SUMMARY:
According to randomized controlled trial requirement, the therapeutic effectiveness of cooled-probe microwave ablation and radiofrequency ablation on early-stage hepatocellular carcinoma is compared to find a better approach for minimally invasive thermal ablation.

DETAILED DESCRIPTION:
According to following enrollment standard, about >400 cases of biopsy-proved hepatocellular carcinoma(HCC) patients will be involved in the study. They will be treated with percutaneously microwave ablation (MWA) and radiofrequency ablation(RFA). The indications of patients enrolled in the study were as follows: tumor size ≤5cm in diameter, tumor number ≤3, Child-Pugh class A or B classification, no evidence of extrahepatic metastasis, vein or bile duct tumor embolus, and no any other anti-cancer treatment was accepted. MWA or RFA is selected for the patient according to the sequence of their visit to the hospital based on randomization number arrangement produced by SPSS 16.0 statistical software. The therapeutic effectiveness will be compared between two modalities.

ELIGIBILITY:
Inclusion Criteria:

* tumor size ≤5cm in diameter,
* tumor number ≤3,
* Child-Pugh class A or B classification,
* no evidence of extrahepatic metastasis,
* vein or bile duct tumor embolus, and
* no any other anti-cancer treatment

Exclusion Criteria:

* not meeting the inclusion criteria

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2008-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cumulative survival rates were calculated by the Kaplan-Meier method, and comparison between MWA and RFA was done by the log-rank test. | up to 79 months

SECONDARY OUTCOMES:
disease free survival rates were calculated by the Kaplan-Meier method, and comparison between MWA and RFA was done by the log-rank test. | up to 79 months
Local tumor progress rates were calculated by the Kaplan-Meier method, and comparison between MWA and RFA was done by the log-rank test. | up to 79 months
An independent Student's t-test was used for comparing treatment parameters(power, time, session,etc)between MWA and RFA. | up to 79 months
Wilcoxon test was used for comparing liver function between MWA and RFA. | up to 79 months

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China